CLINICAL TRIAL: NCT04886817
Title: A Health Systems Intervention to Reduce Sugar-Sweetened Beverage Consumption in Young Children and Families
Brief Title: Intervention to Reduce Sugar-Sweetened Beverage (SSB) Consumption in Children and Families
Acronym: SCOPE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00062659
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff collecting data on the primary outcome of beverage consumption at 3 and 6 month follow-up will be blinded to group allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group participants in this study will not receive any intervention as is the current standard of clinical care for excess sugary drink consumption. They will receive monthly check-in reminders from research staff to promote engagement and retention and will participate in data collection visits at baseline, 3 and 6 months.
- Intervention (Experimental): Intervention group participants will receive a 6-month behavioral intervention with the following components:
  1. A water promotion toolkit that includes water bottles, water flavor infusers, stickers to decorate bottles, and a children's book about water consumption, as well as instructions for other intervention components (how to view video, download app, and prepare for calls)
  2. A 5-minute educational video that introduces parents to healthy drink choices for the family.
  3. Ready, Set Gulp! A smartphone application for families that will help all family members track their beverage intake, find out how much water and sugar they are consuming, set goals, compete for points, answer quiz questions and create new recipes for flavor infused water.
  4. A series of 14 interactive voice response phone calls to parents over 6 months that educate parents on topics relevant to improving family drink choices.
  Interventions: Behavioral: Pilot Intervention to reduce SSB consumption in children and families

INTERVENTIONS:
Behavioral: Pilot Intervention to reduce SSB consumption in children and families — A 6-month intervention based on the use of 4 components: an educational video, provision of a water-promotion "toolkit," a mobile phone application (app), and a series of 14 computerized interactive voice response (IVR) phone calls to parents to compare families' SSB's consumption behaviors
  Arms: Intervention

SUMMARY:
Pilot randomized trial of a technology-based intervention to reduce sugary drink consumption and promote water intake in families with young children.

DETAILED DESCRIPTION:
This is a pilot 2-arm randomized trial among 60 families of 1-8 year old children who currently over-consume sugary drinks. The study team will randomize families to either an intervention group, that will receive a behavioral intervention consisting of an educational video, water promotion toolkit, mobile phone app, and series of educational phone calls, or to a control group that will not receive this intervention. The study team will compare 6-month change in child and parental beverage consumption between groups. Exploratory analyses will examine child weight (kg) and Body Mass Index (BMI) z-score (BMIz) outcomes, and compare intervention effects across race/ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Child 1-8 years old who receives health care attention at Wake Forest pediatric or family medicine practices
* Child consumes 2 or more SSB and/or fruit juice total per day
* Child with no chronic health condition
* Child has not seen nutritionist or visited our family-based weight management clinic in the past year
* parent/caregiver who has not watch educational video "Get in the Zero Zone"
* parent/caregiver has a smartphone and reliable internet
* parent/caregiver able to communicate well in English

Exclusion Criteria:

* Child doesn't meet age criteria
* Child consumes less than 2 SSB and/or fruit juice total per day
* Child with a chronic health condition
* Child has seen nutritionist or visited our family-based weight management clinic in the past year
* parent/caregiver has watched educational video "Get in the Zero Zone"
* parent/caregiver has completed interview or usability test
* parent/caregiver doesn't have a smartphone or reliable internet
* parent/caregiver not able to communicate well in English

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Change in child sugary drink serving consumption | from baseline to month 3
  change in a child's combined consumption of Sugar-Sweetened Beverages (SSB)+Fruit Juice (FJ), measured as total servings per day, at 3 months after starting intervention, measured with Beverage Intake Questionnaire (BevQ15) instrument
Change in child sugary drink serving consumption | from baseline to month 6
  change in a child's combined consumption of Sugar-Sweetened Beverages (SSB)+Fruit Juice (FJ), measured as total servings per day, at 6 months after starting intervention, measured with Beverage Intake Questionnaire (BevQ15) instrument

SECONDARY OUTCOMES:
BevQ 15 - Children Change in Servings of Beverages | from baseline to month 3, from baseline to month 6
  changes in total servings children including water and unsweetened milk
BevQ 15 - Children Change in total Volume of Beverages | from baseline to month 3, from baseline to month 6
  changes in total volume of beverages consumed by children including water and unsweetened milk
BevQ 15 - Children Change in total calories of beverages consumption | from baseline to month 3, from baseline to month 6
  Changes in calories of beverages consumed by children including water and unsweetened milk
BevQ 15 -Parental Change in Sugary beverage consumption | from baseline to month 3, from baseline to month 6
  changes in parental beverage consumption sugary drink serving
BevQ 15 -Parental Change in Beverage Consumption | from baseline to month 3, from baseline to month 6
  changes in total servings for parents including water and unsweetened milk
BevQ 15 -Parental Change in Volume of Beverage Consumption | from baseline to month 3, from baseline to month 6
  changes in total volume for parents including water and unsweetened milk
BevQ 15-Parental Change in Calories of Beverage Consumption | from baseline to month 3, from baseline to month 6
  changes in total beverage calories for parents including water and unsweetened milk
Changes in parent knowledge | from baseline to month 3, from baseline to month 6
  Survey knowledge items will be "scored" in terms of correct or not with a range of 0-17 possible points, with higher score demonstrating more knowledge about SSB and FJ, including how SSB are related to possible health consequences and perceived healthfulness of different beverages.
Changes in Parent Attitudes | from baseline to month 3, from baseline to month 6
  Attitude and belief items will be reported individually, as these are not objectively correct or incorrect and represent a subjective state of the parent's point of view. These will be reported out as frequencies / descriptive statistics, with change in proportion responding a certain way examined over follow-up. Statistician will use Statistical Analysis Software (SAS) for quantifying qualitative data.
Changes in Parent Beliefs | from baseline to month 3, from baseline to month 6
  Belief items will be reported individually, as these are not objectively correct or incorrect and represent a subjective state of the parent's point of view. These will be reported out as frequencies / descriptive statistics, with change in proportion responding a certain way examined over follow-up. Statistician will use Statistical Analysis Software (SAS) for quantifying qualitative data.
Child Weight Change | from baseline to month 3, from baseline to month 6
  change in child weight (kg) using Electronic Health Record (EHR) data
Child Body Mass Index Z-Score (BMIz) Change | from baseline to month 3, from baseline to month 6
  change in child BMIz also using EHR data

OTHER OUTCOMES:
Single Item Literacy Screener (SILS) | baseline
  The SILS is a single item question intended to identify adults in need of help with printed health material. The SILS asks, "How often do you need to have someone help you when you read instructions, pamphlets, or other written material from your doctor or pharmacy?" Possible responses are 1-Never, 2-Rarely, 3-Sometimes, 4-Often, and 5-Always
Modified Version of the Mobile Device Proficiency Questionnaire (MDPQ) | baseline
  This questionnaire asks about the ability to perform a number of tasks with a mobile device. The MDPQ asks seniors to select how easily they could perform 19 mobile device skills from Not at all, Not very easily, Somewhat easily, or very easily.
NCI's 26-item Dietary Screener Questionnaire (DSQ) | baseline, month 6
  The study team will use only 19 items of the DSQ to assess intake of fruits and vegetables, whole grains, added sugars, dairy, fiber, and calcium. DSQ will be asked of parent, responding for child and will exclude questions about beverages as those would be redundant to questions already included in the Bevq-15 instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina H Lewis, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT04886817/ICF_000.pdf